CLINICAL TRIAL: NCT01011296
Title: A Randomized, Placebo Controlled, Double-Blind, Third Party Open, Parallel Group, First In Human Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04427429 Administered Intravenously To Healthy Adult Volunteers
Brief Title: First In Human Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04427429 Administered Intravenously To Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B0141001
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single IV Dose 1 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 2 (Experimental)
  Interventions: Drug: PF-04427429
- Single IV Dose 3 (Experimental)
  Interventions: Drug: PF-04427429

INTERVENTIONS:
Drug: PF-04427429 — Single 0.2mg dose of intravenous infusion
  Arms: Single IV Dose 1
Drug: PF-04427429 — Single 1mg dose of intravenous infusion
  Arms: Single IV Dose 2
Drug: PF-04427429 — Single 3 mg dose of intravenous infusion
  Arms: Single IV Dose 3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-04427429 administered intravenously to healthy adult volunteers.

DETAILED DESCRIPTION:
Phase 1 clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 50 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight of between 50 kg and 100 kg inclusive.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Willing and able to comply with the requirement for using the recommended highly effective contraceptive methods throughout the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, genitourinary, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, symptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of febrile illness within 5 days prior to the first dose.
* A positive urine drug screen

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety (incidence/severity of adverse events and clinical laboratory abnormalities, mean change from baseline/placebo in vital signs/body temperature, mean change from baseline in 12 lead electrocardiogram parameters compared to baseline/ placebo) | anticipated time is up to 84 days post dose
Safety continued (categorical summary of QTcF compared to baseline between dose groups and placebo, concentration QTcF relationship, ADA responses, IV injection site reactions) | anticipated time is up to 84 days post dose to 84 days
Pharmacokinetics (Free plasma concentrations of PF-04427429 will be measured by a validated assay and non-compartmental PK parameters will be determined for each dose) | anticipated time is up to 84 days post dose days

SECONDARY OUTCOMES:
Pharmacodynamics (free and total CGRP plasma concentrations will be measured, the PK-PD relationship between plasma PF-04427429 concentrations and free/total CGRP concentrations will be characterized) | anticipated time is up to 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Phoenix, Arizona, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0141001&StudyName=A%20Randomized%2C%20Placebo%20Controlled%2C%20Double-Blind%2C%20Third%20Party%20Open%2C%20Parallel%20Group%2C%20First%20In%20Human%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20PF-04427429%20Administered%20Intravenously%20To%20Healthy%20Adult%20Volunteers